CLINICAL TRIAL: NCT01331876
Title: Evaluation and Comparison of Cerebral Activities Modifications Associated With Two Different Cognitive and Behavioral Therapies for Obsessive Compulsive Disorder Patients
Brief Title: Modification of Cerebral Activity of Obsessive Compulsive Disorder (OCD) Patients During Cognitive and Behavioral Therapy
Acronym: TOC TOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C09-02; 2009-A00652-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-03-29; First posted 2011-04-08 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2012-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Cognitive and Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- reference therapy (Experimental): 20 OCD patients following 15 sessions of the reference CBT (Bouvard,2006)
  Interventions: Behavioral: Cognitive and behavioral Therapy
- experimental therapy (Experimental): 20 OCD patients following 15 sessions of reference CBT associated with a new psychopedagogic task developed by our team.
  Interventions: Behavioral: Cognitive and behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive and behavioral Therapy — 15 CBT sessions with a psychologist expert in OCD treatment

SUMMARY:
Obsessive compulsive Disorder (OCD) is a frequent psychiatric disorder. Obsessions and compulsions are the two manifestations of this disease. Obsessions are recurrent anxious ideas, and compulsions repetitive behavior aiming to decrease this anxiety.

OCD symptoms have been associated with cortical and sub-cortical dysfunctions and more precisely an hyperactivity of prefrontal cortex / basal ganglia loops.

Functional neuro-imagery studies have shown a significant decrease of orbito-frontal cortex, anterior cingulate cortex, caudate nucleus and cerebellum activities after two OCD reference treatments : medication and Cognitive and Behavioral Therapy (CBT).

Two groups of 20 patients are included in this study and follow a CBT for 15 sessions. They are randomised in two groups : one proposing a "reference CBT", the other associate CBT to a new psychopedagogic task developed by the investigators team.

Clinical investigations and neuro-imagery data are collected at the main steps of therapies : before, during (half-therapy), at the end of therapies and 6 month later. Symptoms severity, patients and relatives quality of life are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65;
* Following Obsessive Compulsive Disorder criteria according to DSM IV(300.3 ;MINI 5.0.0);
* OCD severity range from 20 to 30 on the Y-Brown obsessive compulsive scale;
* Having checking symptoms;
* Understanding and accepting the study;
* Giving his written informed consent to the study.

Exclusion Criteria:

* Claustrophobia;
* Cerebral abnormality;
* Chronic absenteism to CBT (more than 5 missed sessions during the whole therapy).

In case of exclusion of the study either decided by the patient himself or by the investigator, a debriefing is proposed by a psychologist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Changes in brain activity associated with different types of Cognitive Behavioral Therapy Obsessive Compulsive Disorder | before CBT, at half CBT (1.5 month), after CBT (3 months) and 6 six months later
  Evaluation and comparison of changes in brain activity associated with different types of Cognitive Behavioral Therapy in patients with Obsessive Compulsive Disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpêtrière hospital, Paris, France

REFERENCES:
- [Background] Haynes WIA, Clair AH, Fernandez-Vidal S, Gholipour B, Morgieve M, Mallet L. Altered anatomical connections of associative and limbic cortico-basal-ganglia circuits in obsessive-compulsive disorder. Eur Psychiatry. 2018 Jun;51:1-8. doi: 10.1016/j.eurpsy.2018.01.005. Epub 2018 Mar 4. PMID 29514116